CLINICAL TRIAL: NCT00167167
Title: Treatment of Relapsed Leukemia After Allogeneic Bone Marrow Transplantation Using Donor-derived Lymphocytes
Brief Title: Donor Lymphocyte Infusion (DLI) for Relapsed (Post Transplant) Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Jeffrey Miller, MD, Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9510M10277; MT1995-24; 1996LS146
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Leukemia, Myeloid, Chronic; AML; MDS; Leukemia, Lymphocytic, Acute
Keywords: Donor Lymphocyte Infusion; relapse; post-transplant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMT patients (Experimental): All patients treated.
  Interventions: Procedure: Donor Lymphocyte Infusion

INTERVENTIONS:
Procedure: Donor Lymphocyte Infusion — Certain immune cells in your donor's blood called "lymphocytes" have been shown to fight cancer after bone marrow transplantation. We plan to transfuse large numbers of donor's "lymphocytes" in the hope of activating the recipient's immune system to attack cancer.

SUMMARY:
In this study our hypothesis is that infusion of donor lymphocyte immune cells from the subject's bone marrow donor will activate the subject's immune system to attack their cancer.

DETAILED DESCRIPTION:
We will collect immune cells or lymphocytes from the donor's blood using a cell separator. The blood lymphocytes will be given to the subjects through a catheter. If the subjects have no complications of the first course of infusions, we may decide to give them "lymphocytes" aa second time while subjects are in remission in an attempt to prevent their disease from relapsing. A bone marrow test will be taken prior to infusion of lymphocytes as part of the clinical evaluation to receive this treatment. After lymphocyte infusions, a bone marrow will be examined about every three months for the first year to monitor progress from this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CML, AML, MDS or ALL relapsed after related or unrelated donor allogeneic marrow transplantation.
* Patients must be within one year of identification of relapse or if beyond that time period, must have some evidence of donor DNA by RFLP or cytogenetics.
* Patients may have evidence of relapse based on molecular, cytogenetic or morphologic criteria.
* CML patients must have cytogenetic evidence of relapse or if Ph negative to start, obvious evidence of relapse other than minimal residual disease.
* Patients must have <30% marrow blasts on a marrow biopsy performed within two weeks of the first donor lymphocyte infusion.
* Patients with >30% blasts can become eligible for donor lymphocytes after reinduction with any standard therapy regimen.
* Patients with AML, MDS or ALL achieving a CR with standard therapy regimens are eligible for this protocol.
* Patients who relapse with their initial disease or develop a second malignancy after related or unrelated donor allogeneic marrow transplantation with other initial diagnoses (such as but not limited to CLL, lymphoma, myeloma, juvenile CML, sarcoma, breast cancer) may also be included in this protocol. Patients will be eligible with or without other adjunct chemotherapy or radiation therapy. Post-transplant lymphomas (often referred to as EBV-associated lymphomas) will be eligible for donor leukocyte infusions on this protocol. Treatment with donor leukocytes under this protocol is restricted to malignant diseases only. Graft failure or relapse of non-malignant disorders is excluded from receiving donor leukocyte infusions on this protocol. Autologous transplant patients who relapse are not eligible for this protocol. Patients with malignant diseases amenable to other curative therapy are not eligible (i.e. skin cancers).

Exclusion Criteria:

* Patients with concurrent signs of acute or chronic graft-versus-host disease requiring ongoing treatment at the time of relapse will be ineligible.
* Patients with >30% marrow blasts at the time of therapy will be ineligible.
* Patients on prednisone, cyclosporine, Imuran or other immunosuppressive medications are not eligible until these medications are discontinued for at least 2 weeks without a flare of GVHD.
* CML patients in complete cytogenetic remission who are bcr/abl positive by PCR only are not eligible.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 1995-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Freedom of Disease: Bone marrow histology, cytogenetic analysis and RFLP will be studied. Data will be collected and tabulated. | before, at 3 months, 6 months, 9 months and 12 months after donor lymphocyte infusions

SECONDARY OUTCOMES:
Toxicity | during the infusion and immediately thereafter
All data concerning acute toxicity including allergic reactions, capillary leak syndrome, and other Grade 4 toxicity will be collected and tabulated. | during the infusion,immediately thereafter, and at 1 month, 3 months, 6 months, 9 months, 1 year and yearly.
Graft-versus-host disease will be staged using criteria routinely used in allogeneic bone marrow transplant settings and will be tabulated. | ongoing
Marrow Aplasia including duration, treatment and outcomes. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — University of Minnesota Medical Center
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States